CLINICAL TRIAL: NCT00997958
Title: Phase I Study of CellCept for Advanced Pancreatic Cancer
Brief Title: Study of CellCept for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Robert L. Fine, Associate Professor of Hematology and Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA1127
Record Dates: First submitted 2009-10-14; First posted 2009-10-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CellCept (Experimental): Administered in tablet form twice daily one hour after eating.
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Mycophenolate mofetil — Dose escalation increasing successively from 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, and 5.0 grams p.o. bid.
  Each patient will be treated for eight weeks (56 days).

SUMMARY:
Mycophenolate Mofetil (CellCept) is an FDA approved, well tolerated, oral medication used to prevent the body's immune system from attacking transplanted organs. It has never been studied in patients with pancreatic cancer but some preliminary studies have shown that it may antagonize tumor growth. The goals of this study are to find out how much of this drug can safely be taken by patients with advanced pancreatic cancer and to assess the variation of the level of the drug in the blood. Patients will take the drug twice a day at a given dose and the safety of the drug will be monitored through patient symptoms and blood tests. The disease burden will be assessed by radiographic studies at the beginning and end of the study. The patient will take the drug for a total of eight weeks.

DETAILED DESCRIPTION:
Mycophenolate Mofetil (CellCept) is a prodrug whose active metabolite, mycophenolic acid (MPA), acts as an immune suppressant by inhibiting de novo guanosine synthesis. CellCept is FDA approved to prevent rejection of transplanted organs. It is well tolerated, orally dosed, and has some known antitumor effects. It has never been studied in pancreatic cancer and the maximum tolerated dose is not known. In vitro studies in our lab with human pancreatic cancer lines found that MPA was a potent inhibitor of pancreatic cancer cell growth and induced apoptosis. The objectives of this study are to identify the maximum tolerated dose of CellCept in patients with advanced pancreatic cancer that have failed at least two prior chemotherapy regimens and assess its pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of pancreas.
* Disease stage IV, locally advanced and/or metastatic.
* Measurable disease: Any mass reproducibly measurable in two perpendicular diameters by x-ray, physical examination, CT or MRI scan.
* The following lesions conventionally are not considered measurable:

  * CNS lesions
  * Blastic or lytic bone lesions (which will be documented and followed)
  * Radiated lesions unless progression after RT is documented
* Ineligible for other high priority national or institutional studies.
* Prior therapy allowed:

  * Chemotherapy (at least one prior regimen)
  * > 3 weeks since last chemotherapy
  * > 3 weeks since surgery
  * ≥ 4 weeks since RT
* Non pregnant, non lactating women with a negative serum α-HCG test within one week of starting the study, AND
* Must be willing to consent to the use of two forms of contraception (at least one barrier) if of childbearing potential while on trial and six weeks after CellCept has been stopped.
* Clinical Parameters:

  * Life expectancy ≥ 3 months
  * Age 18 to 70 years
  * Brain CT or MRI no visible metastases
  * Performance status 0-2 (ECOG- see appendix B)
  * HIV negative or never tested
* Required initial laboratory data:

  * Normal
  * White cell count ≥3000 cells / μl
  * Platelet count ≥100,000 platelets / μl
  * BUN ≤1.5 x normal 20 mg/dl
  * Creatinine ≤1.5 x normal 1.0 mg/dl
  * Total Bilirubin ≤3.0 mg/dl
  * AST, ALT ≤3.0 x normal 38 U/L
  * Alkaline Phosphatase ≤3.0 x normal 96 U/L
  * Albumin ≥2.5 g/dl
* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, adverse effects, risks, and discomforts.
* Prior malignancy in last 5 years: The cancer must be curatively treated carcinoma in situ of the cervix or skin cancer.
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection).
* Absence of concurrent treatment with cholestyramine, acyclovir, cyclosporine, or antacids with magnesium or aluminum hydroxides because of their effects on drug metabolism and serum levels of MPA.
* Absence of active serious digestive system disease as defined at the discretion of the Principal Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-06; Primary Completion 2007-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Identification of maximum tolerated dose of CellCept in patients with advanced pancreatic cancer | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Fine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States